CLINICAL TRIAL: NCT07249580
Title: A Comparative Study of Self-Efficacy and Perceived Stress Among Physiotherapy Interns in Turkey and Egypt
Brief Title: Comparative Study of Self-Efficacy and Perceived Stress Among Physiotherapy Interns in Turkey and Egypt
Acronym: SEPS-PT
Status: Not yet recruiting | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Mosaab Hassan Ibrahim, M.Sc. Student, Department of Physiotherapy and Rehabilitation, Medipol University
Other Study IDs: E-10840098-202.3.02-3979; E-10840098-202.3.02-3979 (Other: Istanbul Medipol University Non-Interventional Clinical Research Ethics Committee)
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Self-efficacy and Perceived Stress Among Physiotherapy Interns in Clinical Training
Keywords: Physiotherapy Education; Clinical Internship; Self-Efficacy; Perceived Stress; Physiotherapy Students

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Physiotherapy Interns in Turkey: Physiotherapy students from accredited universities in Turkey who are currently completing supervised clinical internships, regardless of academic year. Participants will complete an online questionnaire that includes demographic information, the Physiotherapy Intern Self-Efficacy Scale - Likert Version (PISE-L), and the Perceived Stress Scale (PSS). Responses will be used to evaluate levels of self-efficacy and perceived stress and compared with Egyptian participants.
  Interventions: Other: Online Questionnaire
- Physiotherapy Interns in Egypt: Physiotherapy students from accredited universities in Egypt who are currently engaged in supervised clinical internships, regardless of academic year. Participants will complete the same online survey consisting of demographic questions, the PISE-L, and the PSS. Data will be compared with Turkish interns to assess variations in self-efficacy and perceived stress between the two educational systems.
  Interventions: Other: Online Questionnaire

INTERVENTIONS:
Other: Online Questionnaire — Participants will complete an online self-administered survey consisting of demographic questions, the Physiotherapy Intern Self-Efficacy Scale - Likert Version (PISE-L), and the Perceived Stress Scale (PSS). The questionnaire is used solely for data collection; no behavioral or clinical intervention is applied.

SUMMARY:
This cross-sectional comparative study aims to assess and compare the self-efficacy and perceived stress levels among physiotherapy interns in Turkey and Egypt. The transition from academic study to clinical practice is a critical and often challenging stage for physiotherapy students, requiring the integration of theoretical knowledge and practical skills in real-world clinical environments.

Self-efficacy, derived from Bandura's Social Cognitive Theory, refers to an individual's confidence in their ability to perform specific tasks and achieve desired outcomes. In physiotherapy education, self-efficacy influences clinical reasoning, patient assessment, treatment planning, communication, and interprofessional collaboration. Meanwhile, perceived stress reflects how individuals appraise situations as stressful or demanding, which can affect their confidence and clinical performance.

The study will include 200 physiotherapy interns-100 from Turkey and 100 from Egypt-who are currently completing supervised clinical internships at accredited universities. Data will be collected using an online survey containing three parts: a demographic and educational background form, the Physiotherapy Intern Self-Efficacy Scale - Likert Version (PISE-L), and the Perceived Stress Scale (PSS).

The primary objective is to compare self-efficacy levels between interns from the two countries and explore how differences in educational structures and clinical training environments relate to professional confidence and stress levels. The study also aims to identify correlations between perceived stress and self-efficacy among interns.

Findings from this research are expected to provide valuable insights for improving physiotherapy education programs by highlighting factors that influence students' readiness for professional practice.

DETAILED DESCRIPTION:
This study is a cross-sectional, comparative, observational investigation designed to evaluate and compare the levels of self-efficacy and perceived stress among physiotherapy interns in Turkey and Egypt. The study focuses on understanding how differences in clinical education structure, timing of practical exposure, and learning environments influence the professional confidence and stress management of physiotherapy students transitioning into clinical practice.

Background and Rationale

The transition from academic learning to independent clinical practice represents a critical developmental stage for healthcare professionals, particularly physiotherapists. During this phase, students must apply theoretical knowledge and practical skills in real clinical settings, which can often be demanding and stressful. While technical competence is essential, a key factor influencing success in this stage is psychological readiness-specifically, the belief in one's own capability to manage clinical tasks, known as self-efficacy.

Grounded in Bandura's Social Cognitive Theory, self-efficacy reflects confidence in performing specific actions to achieve desired outcomes. In physiotherapy education, high self-efficacy correlates with better clinical reasoning, patient communication, treatment planning, and professional collaboration. Conversely, low self-efficacy can hinder learning and performance.

Perceived stress is another crucial factor that can influence self-efficacy and clinical competence. Elevated stress levels among interns can negatively affect their confidence, decision-making, and patient interactions. Assessing both self-efficacy and perceived stress offers a comprehensive understanding of physiotherapy students' preparedness for professional practice.

Turkey and Egypt have distinct physiotherapy education models. Turkish programs follow a four-year structure with early and progressive clinical exposure, while Egyptian programs typically last five years, with a mandatory one-year clinical internship after graduation. These structural differences may result in varying levels of clinical confidence and stress among interns. This study aims to explore how these educational variations impact self-efficacy and perceived stress.

Study Objectives

To compare self-efficacy levels between physiotherapy interns in Turkey and Egypt.

To compare perceived stress levels between physiotherapy interns in both countries.

To explore the relationship between perceived stress and self-efficacy.

To identify how differences in educational structures influence professional confidence.

Hypotheses:

H1: Physiotherapy interns in Turkey will report significantly higher self-efficacy scores than those in Egypt.

H2: Physiotherapy interns in Turkey will report significantly lower perceived stress scores than those in Egypt.

Study Design

The study will employ a cross-sectional observational model. Data will be collected through an online survey distributed to physiotherapy interns currently enrolled in accredited universities in Turkey and Egypt.

Participants:

A total of 200 participants (100 from Turkey and 100 from Egypt) will be recruited. Eligible participants must be final-year physiotherapy students currently completing a supervised clinical internship.

Inclusion Criteria:

Currently engaged in a supervised clinical internship.

Sufficient fluency in Turkish or English (depending on the questionnaire language).

Provided informed consent to participate.

Exclusion Criteria:

Already graduated or licensed physiotherapists.

Incomplete responses exceeding 10% of questionnaire items.

Data Collection Instruments

Demographic and Educational Background Form - collects information such as age, gender, university, program type (public/private), total clinical hours, timing of first patient contact, prior healthcare experience, and GPA.

Physiotherapy Intern Self-Efficacy Scale - Likert Version (PISE-L) - a validated 30-item instrument assessing self-efficacy across five domains: clinical reasoning, patient assessment, treatment planning, patient education and communication, and interprofessional collaboration.

Perceived Stress Scale (PSS-10) - a 10-item validated measure assessing individuals' perceived stress over the previous month.

The Turkish version of both scales will be used for Turkish participants, and the English version for Egyptian participants. The translation followed standard forward-backward translation and expert validation procedures to ensure linguistic and conceptual equivalence.

Statistical Analysis

Data will be analyzed using SPSS version 23. Descriptive statistics (mean, standard deviation, frequency, percentage) will summarize participant characteristics. Normality of data distribution will be assessed. Independent t-tests or Mann-Whitney U tests will be used for between-group comparisons depending on data distribution. Correlation analysis will explore relationships between self-efficacy and perceived stress. Significance will be set at p < 0.05.

Ethical Considerations

Ethical approval was obtained from Istanbul Medipol University Non-Interventional Clinical Research Ethics Committee (Decision No. E-10840098-202.3.02-3979, dated June 19, 2025). Participation in the study is voluntary. Informed consent will be obtained electronically before data collection. All data will remain anonymous and confidential, and participants may withdraw at any time without penalty. No personal or identifying information will be collected.

Expected Outcomes

It is anticipated that Turkish physiotherapy interns will demonstrate higher self-efficacy and lower perceived stress levels compared to Egyptian interns, reflecting the differences in educational models and clinical exposure timing. The results are expected to provide insights into optimizing physiotherapy curricula to enhance students' confidence and readiness for clinical practice in both countries.

Significance

The findings will contribute to the body of knowledge on physiotherapy education by identifying key factors that shape clinical preparedness. This research may guide curriculum developers, educators, and policymakers in designing interventions that promote psychological readiness and reduce stress among physiotherapy students worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Physiotherapy students or interns currently enrolled in accredited universities in Turkey or Egypt.
* Actively participating in a supervised clinical internship or practical training at the time of the study.
* Aged between 18 and 30 years.
* Able to read and understand the survey language (Turkish or English).
* Willing to provide informed consent and complete the online questionnaire.

Exclusion Criteria:

* Individuals who have already graduated and are no longer in an internship program.
* Participants with incomplete or invalid survey responses (more than 10% of items unanswered).
* Students who are not currently engaged in any form of clinical internship or practical training.
* Participants who withdraw consent or choose not to complete the survey.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of physiotherapy students from accredited universities in Turkey and Egypt who are currently participating in supervised clinical internships. Participants may be in different academic years, provided they are actively involved in patient care or clinical training as part of their curriculum. All participants will voluntarily complete an online questionnaire in Turkish or English that includes demographic information, the Physiotherapy Intern Self-Efficacy Scale - Likert Version (PISE-L), and the Perceived Stress Scale (PSS).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-Efficacy Level | At the time of survey completion (Baseline)
  The level of self-efficacy among physiotherapy interns will be assessed using the Physiotherapy Intern Self-Efficacy Scale - Likert Version (PISE-L). This scale evaluates confidence across multiple domains including patient assessment, clinical reasoning, treatment planning, communication, and collaboration. The total score reflects the intern's perceived self-efficacy in clinical practice.

SECONDARY OUTCOMES:
Perceived Stress Level | At the time of survey completion (Baseline)
  The perceived stress level among physiotherapy interns will be evaluated using the Perceived Stress Scale (PSS-10), which measures the degree to which situations in life are appraised as stressful. The total score indicates the participant's perceived stress level, with higher scores representing greater perceived stress.

OTHER OUTCOMES:
Relationship Between Self-Efficacy and Perceived Stress | At the time of survey completion (Baseline)
  The relationship between self-efficacy (measured by the Physiotherapy Intern Self-Efficacy Scale - Likert Version) and perceived stress (measured by the Perceived Stress Scale) will be analyzed using correlation statistics to assess the association between the two variables among physiotherapy interns.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Yilmaz Menek, PhD, Study Director — Medipol University
Locations (1):
- Medipol University, Istanbul, Beykoz/İstanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Lankveld W, Jones A, Brunnekreef JJ, Seeger JPH, Bart Staal J. Assessing physical therapist students' self-efficacy: measurement properties of the Physiotherapist Self-Efficacy (PSE) questionnaire. BMC Med Educ. 2017 Dec 12;17(1):250. doi: 10.1186/s12909-017-1094-x. PMID 29233154
- [Background] Milgate W, Copley J, Hill J. Failing professional practice placements in allied health: What do we understand about the student experience? A scoping review. Adv Health Sci Educ Theory Pract. 2024 Mar;29(1):301-327. doi: 10.1007/s10459-023-10243-w. Epub 2023 Jun 7. PMID 37284962
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- See also: Failing professional practice placements in allied health: What do we understand about the student experience? (Advances in Health Sciences Education, 2024) — https://doi.org/10.1007/s10459-023-10243-w
- See also: Published study describing the validation and measurement properties of the Physiotherapist Self-Efficacy (PSE) questionnaire, conceptually related to the current research on physiotherapy intern self-efficacy and perceived stress. — https://doi.org/10.1186/s12909-017-1094-x
- See also: elf-Efficacy with Telehealth Examination: the Doctor of Physical Therapy Student Perspective (Philippine Journal of Physical Therapy, 2023) — https://doi.org/10.46409/002.udav8455
- See also: Clinical stress and academic self-efficacy in undergraduate nursing students (BMC Nursing, 2025) — https://doi.org/10.1186/s12912-025-02836-0